CLINICAL TRIAL: NCT02702518
Title: A Phase I/II Randomized Placebo-Controlled, Double-Blind, Single-Center, Tolerability and Preliminary Efficacy Clinical Trial of Recombinant Human Deoxyribonuclease (rhDNase) Eye Drops in Patients With Ocular Graft-Vs.-Host Disease
Brief Title: rhDNase Eye Drops in Patients With Ocular Graft-Vs.-Host Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The DSMB committee recommended closing the trial because of the COVID-19 risk in this "at-risk" oGVHD population if they came for study visits.
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Genentech, Inc. (Industry); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Sandeep Jain, MD, Associate Professor of Ophthalmology, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-0372; R01EY024966-01A1 (NIH)
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Ocular Graft vs Host Disease; Dry Eye
Keywords: rhDNase I, Pulmozyme, oGVHD, Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — dornase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhDNase I (Active Comparator): rhDNase I 0.1% eye drops 4 times a day for 8 weeks
  Interventions: Drug: rhDNase I
- Vehicle (Placebo Comparator): Drug vehicle eye drops 4 times a day for 8 weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: rhDNase I — rhDNase I, 0.1% eye drops 4 times a day for 8 weeks
  Other Names: Pulmozyme
  Arms: rhDNase I
Drug: Vehicle — Drug vehicle 4 times a day for 8 weeks
  Other Names: Placebo
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the tolerability and preliminary efficacy of rhDNase I eye drops in patients with ocular Graft-vs.-Host disease (oGVHD).

ELIGIBILITY:
Inclusion Criteria:

* The PI and other members of International Chronic Ocular GVHD Consensus Group have established the consensus diagnostic criteria and classification for chronic ocular GVHD.

Table 1: Severity scale in chronic ocular GVHD

Severity scores (points) Schirmer's test (mm) CFS (points) OSDI (points) Conj (points) 0 >15 0 <13 None

1. 11-15 <2 13-22 Mild/Moderate
2. 6-10 2-3 23-32 Severe
3. ≤5 ≥4 ≥33

CFS; corneal fluorescein staining, OSDI; Ocular Surface Disease Index. Conj; conjunctival injection. Severity classification; Total score (points); (Schirmer's test score+ CFS score+ OSDI score+ Conj injection score) = None;0-4, Mild/Moderate; 5-8, Severe, 9-11.

Table 2: Diagnosis of chronic ocular GVHD None (points) Probable GVHD (points) Definite GVHD (points) Systemic GVHD(-) 0-5 6-7 ≥8 Systemic GVHD(+) 0-3 4-5 ≥6

Based on these criteria (Tables 1 and 2),40 patients with definite ocular GVHD will be enrolled. Additionally, all of the following criteria should be met to be eligible for the study:

* Aged 18 years or older.
* Capable of giving informed consent and does provide informed consent.
* Schirmer I <10
* Corneal/ conjunctival (Rose Bengal) staining ≥1
* Ocular symptoms must be considered as annoying or activity limiting (OSDI ≥13; mild).
* Women must be post-menopausal ≥ 1 year, or surgically sterilized. If not, a negative urine pregnancy test is required within 14 days of receiving her first dose of test medication (placebo/ study drug) along with definite evidence of contraceptive use during the duration of the study. Women of reproductive age should use a method of birth control that is acceptable to the subject and the study doctor. This may include oral contraceptive pills, birth control implants, barrier methods or abstinence. If a subject mentions she suspects she may be pregnant after being enrolled, another pregnancy test will be administered. If the test is positive, she will be discontinued from the study immediately.

Exclusion Criteria:

* Subjects will not be eligible for the study if any of the following criteria are met:

  * Allergic to rhDNase I or any similar products, or recipient of rhDNase I eye drops 0.1%.
  * Receiving or have received within 30 days any experimental systemic medication.
  * Active ocular infection or ocular allergies.
  * Any history of eyelid surgery or ocular surgery within the past 3 months.
  * Corneal epithelial defect larger than 1 mm2 in either eye.
  * Have active drug/alcohol dependence or abuse history.
  * Vulnerable populations, such as neonates, pregnant women, children, prisoners, institutionalized individuals, or others who may be considered vulnerable populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-04; Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Jain, MD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - Translational Clinic of Corneal Neurobiology laboratory, Illinois Eye and Ear Infirmary, University of Illinois at Chicago, Chicago, Illinois
  - University of Illinois Eye and Ear Infirmary, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tibrewal S, Sarkar J, Jassim SH, Gandhi S, Sonawane S, Chaudhary S, Byun YS, Ivanir Y, Hallak J, Horner JH, Newcomb M, Jain S. Tear fluid extracellular DNA: diagnostic and therapeutic implications in dry eye disease. Invest Ophthalmol Vis Sci. 2013 Dec 11;54(13):8051-61. doi: 10.1167/iovs.13-12844. PMID 24255046
- [Result] Sonawane S, Khanolkar V, Namavari A, Chaudhary S, Gandhi S, Tibrewal S, Jassim SH, Shaheen B, Hallak J, Horner JH, Newcomb M, Sarkar J, Jain S. Ocular surface extracellular DNA and nuclease activity imbalance: a new paradigm for inflammation in dry eye disease. Invest Ophthalmol Vis Sci. 2012 Dec 17;53(13):8253-63. doi: 10.1167/iovs.12-10430. PMID 23169882
- [Derived] Mun CS, Surenkhuu B, Chen YF, Atassi N, Mun J, Kim C, Sheth T, Sarwar MA, Pradeep A, Jain S. Recombinant Deoxyribonuclease I Eye Drops for Ocular Graft Versus Host Disease: Results of a Randomized Clinical Trial. Eye Contact Lens. 2024 May 1;50(5):233-240. doi: 10.1097/ICL.0000000000001078. Epub 2024 Feb 23. PMID 38407974
- See also: Principal Investigator description — https://hospital.uillinois.edu/find-a-doctor/sandeep-jain
- See also: Description of research laboratory — http://cornealneurobiology.uic.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rhDNase I | Vehicle
Started | 29 | 29
Completed | 26 | 25
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rhDNase I | Vehicle | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [46 to 60] | 52 [44 to 60] | 53 [44 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 18 | 20 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 24 | 23 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58
Indication (%) [Count of Participants; unit: Participants]
  Leukemia | 20 | 21 | 41
  Lymphoma | 3 | 1 | 4
  Multiple myeloma | 4 | 1 | 5
  Myeloproliferative disorders | 1 | 1 | 2
  Other | 1 | 5 | 6
BMT date (years) [Median (Inter-Quartile Range); unit: years] | 5.2 [1.9 to 9.5] | 2.2 [1.2 to 3.6] | 2.8 [1.3 to 6.5]
Heart rate [Median (Inter-Quartile Range); unit: Beats per minute (BPM)] | 84 [69.8 to 88.2] | 81 [73 to 88] | 83.5 [70.25 to 88]
Temperature [Median (Inter-Quartile Range); unit: degrees Fahrenheit] | 97.8 [97.4 to 98] | 97.6 [96.9 to 98] | 97.7 [97.13 to 98]
Systemic GVHD [Number; unit: participants] — Population: These counts only correspond to subjects with systemic GVHD. Some subjects had more than one presentation of systemic GVHD.
  participants
    Skin: number analyzed (Participants) | 20 | 21 | 41
    Skin | 13 | 14 | 27
    GI: number analyzed (Participants) | 20 | 21 | 41
    GI | 3 | 3 | 6
    Mouth: number analyzed (Participants) | 20 | 21 | 41
    Mouth | 12 | 12 | 24
    Lung: number analyzed (Participants) | 20 | 21 | 41
    Lung | 3 | 2 | 5
    Joint: number analyzed (Participants) | 20 | 21 | 41
    Joint | 1 | 0 | 1
    Genitalia: number analyzed (Participants) | 20 | 21 | 41
    Genitalia | 3 | 1 | 4
    Other: number analyzed (Participants) | 20 | 21 | 41
    Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Corneal Surface Staining as Measured by Dye Staining Within Groups.
Description: Corneal staining score as measured by dye staining using National Eye Institute (NEI) grading scale. Dye was applied to each eye and a slit lamp was used to observe corneal staining. NEI scale relies on a chart that divides the cornea into 5 sections and assigns a value from 0 (absent) to 3 (severe) to each section, based on the density of punctate staining, final staining score being the sum of individual section scores with a range of 0 (minimum) -15 (maximum) points. Complete corneal staining clearance with dye defined as a score of 0 indicating the best outcome.
Time Frame: Between baseline and at 8 weeks of treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | rhDNase I | Vehicle
Number analyzed (Participants) | 29 | 29
score on a scale
  Week 8 | 3.5 [2.75 to 5.00] | 4.5 [4.00 to 6.00]
  Baseline | 5.00 [3.00 to 7.00] | 4.00 [3.00 to 6.00]
Statistical Analysis 1: Comparison: rhDNase I; For the outcome measure corneal staining, data at week 8 was compared with data at baseline to determine if a change was significant (threshold p < 0.05); Test type: Other; p < 0.001, Mixed Models Analysis — p-values were calculated via linear quantile mixed model for continuous variables with missing data
Statistical Analysis 2: Comparison: Vehicle; For the outcome measure corneal staining data at week 8 was compared with data at baseline to determine significant change; Test type: Other; p = 0.2324, Mixed Models Analysis — p-values were calculated via linear quantile mixed model for continuous variables with missing data

2. Secondary Outcome: The Change in Ocular Surface Disease Index (OSDI) Score Within Groups
Description: Ocular Surface Disease Index (OSDI), a 12-item questionnaire, assesses symptom of ocular irritation in dry eye disease (DED) and how it affects functioning related to vision in the past week. It has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on 0 to 4 scale with 0 being "none of the time" and 4 being "all of the time." OSDI score range from 0-100 with score 0-12 being normal, 13-22 being mild DED, 23-32 being moderate DED, and >33 being severe DED. OSDI=[(sum of scores for questions answered)×100]/[(total questions answered)×4]
Time Frame: Between baseline and at 8 weeks of treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | rhDNase I | Vehicle
Number analyzed (Participants) | 29 | 29
score on a scale
  Week 8 | 18.4 [9.16 to 33.1] | 25.0 [16.5 to 44.3]
  Baseline | 45.5 [31.8 to 50.0] | 37.5 [31.8 to 56.0]
Statistical Analysis 1: Comparison: rhDNase I; For the outcome measure OSDI, data at week 8 was compared with data at baseline to determine if a change was significant (threshold p < 0.05); Test type: Other; p = 0.001, Mixed Models Analysis — p-values were calculated via linear quantile mixed model for continuous variables
Statistical Analysis 2: Comparison: Vehicle; For the outcome measure OSDI data at week 8 was compared with data at baseline to determine significant change; Test type: Other; p = 0.2257, Mixed Models Analysis — p-values were calculated via linear quantile mixed model for continuous variables

ADVERSE EVENTS:
Time Frame: Between baseline and 8-weeks of treatment
Arm/Group | rhDNase I | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 17/29 | 10/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rhDNase I (N=29) | Vehicle (N=29)
Ocular discomfort (Eye disorders) | 6 | 1
Burning sensation (Eye disorders) | 6 | 3
Pain (Eye disorders) | 3 | 2
Blurring of vision (Eye disorders) | 4 | 4
Light sensitivity (Eye disorders) | 4 | 1
Dryness (Eye disorders) | 5 | 4
Redness (Eye disorders) | 3 | 2
Foreign body sensation (Eye disorders) | 4 | 3
Itching (Eye disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT02702518/Prot_SAP_000.pdf